CLINICAL TRIAL: NCT03821077
Title: Prospective Observational Study to Evaluate the Efficacy and Safety of Treatment With "Allergovac Poliplus" in Polysensitized Patients With Allergic Rhinitis/Rhinoconjunctivitis, With or Without Associated Asthma
Brief Title: Study to Evaluate the Efficacy and Safety of "Allergovac Poliplus" in Polysensitized Patients With Allergic Rhinitis/Rhinoconjunctivitis, With or Without Asthma
Acronym: ARES
Status: Completed | Type: Observational
Sponsor: Roxall Medicina España S.A (Industry)
Responsible Party: Sponsor
Other Study IDs: ROX-ALE-2018-01
Record Dates: First submitted 2019-01-24; First posted 2019-01-29 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Rhinitis, Allergic; Rhinoconjunctivitis
Keywords: Allergen immunotherapy (AIT); Rhinitis; Rhinoconjunctivitis; Subcutaneous Immunotherapy (SCIT); Allergovac Poliplus
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis | interventions — Desensitization, Immunologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Allergen Immunotherapy (AIT) — Immunotherapy vaccine with 2 allergenic extracts mixtures (pollens or mites)in polimerized-depot formulation
  Other Names: Allergovac Poliplus

SUMMARY:
This is an observational prospective multicenter clinical study, to evaluate the efficacy and safety of the treatment with Allergovac Poliplus subcutaneous immunotherapy (SCIT) with a mixture of 2 allergenic extracts (pollens or mites), in polymerized-depot formulation, administered in its different available allergenic extracts mixtures (2 pollens or 2 mites), and in one of the 2 recommended administration schedules (1 Day or Rapid).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 5 and 60 years with allergic rhinitis or rhinoconjunctivitis mediated by IgE, caused by sensitization to more than one allergenic source (pollens or mites) and with or without associated mild / moderate asthma.
2. Patients susceptible to receive treatment with Allergovac Poliplus (SCIT), according to usual clinical practice
3. Patients who have given their signed informed consent.

Exclusion Criteria:

1. Patients who have received or initiated treatment with Allergovac Poliplus previously to study inclusion.
2. Patients who have received previous immunotherapy treatment, both subcutaneous (SCIT) and sublingual (SLIT), with any of the allergenic extracts that they plan to receive, in the 5 years prior to study inclusion.
3. Patients who in the opinion of the investigator may present difficulties that prevent the understanding of what was written in the informed consent form or the completion of self-administered questionnaires / scales or the patient's diary.
4. Patients who are participating in another clinical trial or observational study with any drug.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients between 5-60 years, with allergic rhinitis/rhinoconjunctivitis with or without asthma, polisensitized to pollens/mites.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Combined Symptoms and Medication Score (CSMS) | Basal-12 months
  The score ranged from 0 to 6 points and is obtained as follows:
  Symptoms Score (SS) (from 0 to 3 points) + Medication Score (MS) (from 0 to 3 points). Through these 2 sub-scales the total score of the Combined Symptom and Medication Scale (CSMS) is obtained as follows:
  CSMS = SS (0-3) + MS (0-3) = 0-6 points The 0 value indicate no symptoms and no medication, and 6 points indicate the worst state of symptoms and the highest medication step

SECONDARY OUTCOMES:
Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | Basal-12 months
  The RQLQ has 28 questions in 7 domains (activity limitation, sleep problems, nose symptoms, eye symptoms, non-nose/eye symptoms, practical problems and emotional function). It is a self-administered questionnaire where patients respond to each question on a 7-point scale (0 = not impaired at all - 6 = severely impaired). The overall RQLQ score is the mean of all 28 responses and the individual domain scores are the means of the items in those domains. Higher scores reflect lower quality of life.
Total number, percentage, severity and gradation of adverse reactions | Basal- 6 months-12 months
  Total number, percentage, severity and gradation of adverse reactions reported (local and systemics), in relation to the total number of patients and the total administered doses, both globally and according to each administration schedule.
Patient´s Tolerability assessment using a Likert-type scale | 6 months-12 months
  Patient´s Tolerability assessment using a Likert-type scale, with a score of 1 to 4 points (from 1 = I have tolerated it very well to 4 = I have tolerated it very badly)
Patient's perception of the improvement in their global status using a Likert-type scale | 12 months
  Evaluation of the patient's perception of the improvement in the global state of the pathology, using a Likert-type scale, with a score of 1 to 4 points (from 1= good or excellent improvement to 4 = worsening)
Patient's Satisfaction using a Likert scale | 12 months
  Degree of patients' satisfaction with the treatment using a Likert scale, with a score of 1 to 4 points (from 1 = Very Satisfied to 4 = Very dissatisfied)

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Centre Assistencial Baix Llobregat, Cornellà de Llobregat, Barcelona
  - Hospital de Igualada, Igualada, Barcelona
  - GAME Centre Medic, Sant Boi de Llobregat, Barcelona
  - Fundación Hospital Calahorra, Calahorra, La Rioja
  - CAR SAn Millán, Logroño, La Rioja
  - Centro médico Promosalud, Logroño, La Rioja
  - Allercen, Barcelona
  - Centre Medic Catalonia, Barcelona
  - Hospital QuironSalud Barcelona, Barcelona
  - Hospital Sanitas CIMA, Barcelona

IPD SHARING:
Plan to Share IPD: No